CLINICAL TRIAL: NCT04306835
Title: The Impact of Cognitive Behavioral Therapy for Insomnia on CPAP Therapy Use and Drop Outs in Obstructive Sleep Apnea Syndrome Patients With Insomnia.
Brief Title: The Impact of CBT-i on CPAP Therapy Use and Drop Outs in OSAS Patients With Insomnia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 143201836242
Record Dates: First submitted 2020-02-27; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2019-03

CONDITIONS: Insomnia; Obstructive Sleep Apnea; Cognitive Behavioral Therapy; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Apnea, Obstructive | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP + CBT-i (Active Comparator): Patients treated simultaneously with CPAP for their OSAS and cognitive behavioral therapy for their insomnia.
  Interventions: Behavioral: Cognitive behavioural therapy for insomnia
- CPAP only (No Intervention): Patients suffering from OSAS and insomnia, but only treated with CPAP.

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy for insomnia — a technique for treating insomnia without medications
  Arms: CPAP + CBT-i

SUMMARY:
Patients follow the fully standard sleep test according to the normal procedure. This means that they undergo a polysomnography and fill in a questionnaire. If according to the questionnaire, there is insomnia, the patient also receives an intake interview to check whether this is indeed the case. If the patient has both disorders and meets the inclusion and exclusion criteria, they will be asked to sign the informed consent. If the patient agrees, the CPAP-therapy will be started as usual, simultaneously with CGT-i. The latter will last 7 weeks and will cover the following points: psycho-education, sleep restriction and sleep hygiene, cognition, relaxation and relapse prevention. Because of the design of this study (starting CGT-I as soon as possible after the diagnosis of OSAS) and the groups already planned for CBT-I, it is not possible for all participants to participate in group cognitive behavioral therapy, therefore individual sessions were provided for these participants. The patient comes for monitoring at set times.

ELIGIBILITY:
Inclusion Criteria:

* All patients, male and female, with an OSAS diagnosed by full polysomnography and insomnia diagnosed by questionnaires.
* Age between 18 and 75 years
* Dutch as native language

Exclusion Criteria:

* Patients younger than 18 years and older than 75 years
* Patients with a burn-out
* Patients with restless legs
* Pregnant woman
* Patients who work as shift workers
* Patients with severe psychiatric disorder
* Patients who take sleep medication, unless it can be reduced and stopped during cognitive behavior therapy
* Patients with daily alcohol abuse (men > 3 drinks on any day or 14 per week, women > 2 drinks on any day or 7 per week)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
The number of drop-outs in patients participating in the study. | 12 weeks
  Patiënt who don't use there CPAP anymore.
CPAP habituation in patients participating in the study. | 12 weeks
  The speed of CPAP habituation is determined by reading the CPAP device.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided